CLINICAL TRIAL: NCT07151820
Title: Association of Adverse Events in the Real World With Treatment Adjustments, and Burden of AEs in Patients With Chronic Myeloid Leukemia
Brief Title: A Real-world Study About the Impact of Adverse Events (AEs) on Treatment Adjustments, Healthcare Resource Use, and Costs Among Chronic Myeloid Leukemia Patients
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CABL001A0US08
Record Dates: First submitted 2025-08-25; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Leukemia, Chronic Myeloid
Keywords: Tyrosine kinase inhibitor; Adverse events; Treatment adjustment; Healthcare resource use; Healthcare costs
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- First Generation (1G) TKI Cohort: Adult CML patients who received imatinib, a 1G TKI.
- Second Generation (2G) TKI Cohort: Adult CML patients who received the following 2G TKIs: dasatinib, nilotinib, or bosutinib.

SUMMARY:
The aim of this study was to assess the frequency of adverse events (AEs) experienced by chronic myeloid leukemia (CML) patients treated with tyrosine kinase inhibitors (TKIs) and evaluate their impact on treatment adjustments as well as the burden of AEs on healthcare resource use (HRU) and costs.

This study used real-world administrative claims data from the PharMetrics Plus database. AEs of interest were selected based on information obtained from the National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines, Chronic Myeloid Leukemia Version 1. 2024 and clinical inputs. Given the nature of claims data, only AEs of interest that required medical attention (i.e., resulted in a claim record) were captured in this study.

ELIGIBILITY:
Inclusion criteria:

Patients who met all of the following criteria were considered for inclusion:

* Had at least two diagnoses for CML- International Classification of Disease, 10th revision, Clinical Modification (ICD-10-CM) code: C92.1x
* Aged 18 years or older at the time of first CML diagnosis
* Received a 1G or 2G TKI after the first CML diagnosis
* Had continuous health plan enrollment (pharmacy and medical benefits) for at least 6 months before the index date (baseline) and 6 months after the index date

Exclusion criteria:

Patients who met any of the following criteria were excluded:

* Patients had 2 or more diagnoses of gastrointestinal stromal tumor ([GIST], ICD-10: C49.Ax) or chronic myelomonocytic leukemia ([CMML], ICD-10: C93.1x) at any time
* Patients had a hematopoietic stem cell transplantation (HSCT) during the baseline period
* Patients had CML-related chemotherapy treatment for accelerated phase (AP)/blast crisis (BC) during the baseline period
* Patients had medical claims associated with a clinical trial during the baseline period up to the end of the observation period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 2546 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-10-22 (Actual)

PRIMARY OUTCOMES:
Number of Patients With AEs of Interest During the Study Period Among Those Without the Specific Event During the Baseline Period | Up to approximately 7 years and 3 months
  The Study Period spanned from treatment initiation until treatment discontinuation, one day before treatment switch to another CML treatment, end of data availability, end of health plan coverage, or death, whichever came first.
Number of Patients With AEs of Interest Among All Patients During the Study Period | Up to approximately 7 years and 3 months
  The Study Period spanned from treatment initiation until treatment discontinuation, one day before treatment switch to another CML treatment, end of data availability, end of health plan coverage, or death, whichever came first.

SECONDARY OUTCOMES:
Number of Patients With Treatment Adjustments During the Observation Period | Up to approximately 7 years and 3 months
  The Observation Period spanned from treatment initiation to the end of data availability, end of health plan coverage, or death, whichever occurred first.
  Treatment adjustments included:
  * Treatment discontinuation
  * Treatment interruption
  * Switching treatment
  * Dose reduction
Duration of First Treatment Interruption | Up to approximately 7 years and 3 months
Time From TKI Initiation to Treatment Adjustment | Up to approximately 7 years and 3 months
  Treatment adjustments included:
  * Treatment discontinuation
  * Treatment interruption
  * Switching treatment
  * Dose reduction
Number of Patients With AEs of Interest Within 30 Days Before Treatment Adjustment | 6 months
  Treatment adjustments included:
  * Treatment discontinuation
  * Treatment interruption
  * Dose reduction
Number of AEs of Interest Within 30 Days Before Treatment Adjustment | 6 months
  Treatment adjustments included:
  * Treatment discontinuation
  * Treatment interruption
  * Dose reduction
Number of Patients by AE of Interest Experienced Within 30 Days Before Treatment Adjustment | 6 months
  Treatment adjustments included:
  * Treatment discontinuation
  * Treatment interruption
  * Dose reduction
Time Between the Last AE of Interest and Treatment Adjustment | 6 months
  Treatment adjustments included:
  * Treatment discontinuation
  * Treatment interruption
  * Dose reduction
Number of Patients by Last AE of Interest Experienced Before Treatment Adjustment | 6 months
  Treatment adjustments included:
  * Treatment discontinuation
  * Treatment interruption
  * Dose reduction
Number of All-cause Healthcare Visits Per-Patient-Per-Year (PPPY) | 6 months
  Healthcare visits included:
  * Inpatient admissions
  * Emergency department visits
  * Outpatient visits
  * Other visits
Number of Patients With One or More All-cause Healthcare Visits | 6 months
  Healthcare visits included:
  * Inpatient admissions
  * Emergency department visits
  * Outpatient admissions
  * Other visits
Number of All-cause Inpatient Days | 6 months
Number of All-cause Inpatient Days Among Hospitalized Patients | 6 months
All-cause Healthcare Costs PPPY | 6 months
  Healthcare costs included:
  * Total costs
  * Medical costs
  * Inpatient costs
  * Emergency department costs
  * Outpatient costs
  * Other costs
  * Pharmacy costs
Annual Mean Number of Healthcare Visits Associated With AEs of Interest | 6 months
  Healthcare visits included:
  * Inpatient admissions
  * Emergency department visits
  * Outpatient admissions
  * Other visits
Annual Mean Costs of Healthcare Visits Associated With AEs of Interest | 6 months
  Healthcare costs included:
  * Total costs
  * Medical costs
  * Inpatient costs
  * Emergency department costs
  * Outpatient costs
  * Other costs
  * Pharmacy costs

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States